CLINICAL TRIAL: NCT06080048
Title: A Ph I Randomized Double-Blind First-in-Human Single Ascending Dose & Multiple Dose Study to Investigate the Safety Tolerability and Pharmacokinetics of SOR102 in Healthy Adult Participants and Patient Volunteers With Mild to Severe Ulcerative Colitis
Brief Title: A Clinical Trial to Assess the Safety of SOR102 in Healthy Participants and Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sorriso Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SOR102-101
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 3 SOR102 QD (Experimental): SOR102 once a day for 6 weeks SOR102 oral capsules
  Interventions: Drug: SOR102
- Part 3 SOR102 BID (Experimental): SOR102 twice a day for 6 weeks SOR102 oral capsules
  Interventions: Drug: SOR102
- Part 3 Placebo (Placebo Comparator): Placebo for twice a day for 6 weeks Placebo oral capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SOR102 — SOR102 capsules
  Arms: Part 3 SOR102 BID; Part 3 SOR102 QD
Drug: Placebo — Matching placebo capsules
  Arms: Part 3 Placebo

SUMMARY:
SOR102-101 is a Phase 1, 3-part, randomised, double-blind, placebo-controlled, FIH study to determine the safety, tolerability, and PK of single, ascending oral doses (SAD) of SOR102 (Part 1) and multiple oral doses (Part 2) of SOR102 in healthy adult participants, and to assess the safety, tolerability, PK, and biological activity of multiple oral doses of SOR102 in patients with mild to severe UC (Part 3).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or females, of any ethnic origin.
* Established diagnosis of UC by standard criteria for >3 months.
* Disease evaluable by sigmoidoscopy.
* Mildly to severely active UC as determined by central reader in combination with other assessments of disease

Key Exclusion Criteria:

* Any diagnosis of IBD except for UC.
* History of fistula(e), strictures or surgery, known intestinal obstruction, or diagnosis of toxic megacolon.
* Concurrent use of any biologic drug.
* Prior primary efficacy failure or secondary loss of response to more than one biologic or new small molecule therapy (i.e., JAK inhibitors or S1P receptor modulators) indicated for the treatment of UC. This does not include prior discontinuation due to drug intolerance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events following oral dosing | Up to 6 weeks in Part 3 or at the time of study discontinuation
  After multiple oral doses administered BID or QD, number of subjects with AEs in the SOR102 dose level cohorts compared with the oral placebo group

SECONDARY OUTCOMES:
SOR102 concentrations following oral dosing | Up to 6 weeks in Part 3 or at the time of study discontinuation
  To determine the concentration of SOR102 in serum, urine and feces.
Incidence of positive ADAs to SOR102 | Following 6 weeks of study treatment in Part 3 or at the time of study discontinuation
  To assess the incidence of positive ADAs to SOR102.
Incidence of positive neutralizing ADA | Following 6 weeks of study treatment in Part 3 or at the time of study discontinuation
  To assess the incidence of positive neutralizing ADA to SOR102 and its monomers in patients with positive ADA to SOR102.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos C Sattler, MD, Study Director — Sorriso Pharmaceuticals
Locations (2):
- Arensia Exploratory Medicine, Tbilisi, Georgia
- Arensia Exploratory Medicine, Kyiv, Ukraine

REFERENCES:
- [Derived] Jairath V, Danese S, D'Haens GR, Feagan BG, Peyrin-Biroulet L, Sands BE, Gaemers I, Westfall M, Terry AQ, Roberts KJ, Barbat S, Wedel P, Benson JM, Sattler C. Safety and pharmacokinetics of SOR102, an oral bispecific inhibitor of TNF and interleukin-23 in healthy participants and patients with ulcerative colitis: a first-in-human, double-blind, randomised, placebo-controlled, phase 1 trial. Lancet Gastroenterol Hepatol. 2026 Jan;11(1):34-45. doi: 10.1016/S2468-1253(25)00296-1. Epub 2025 Nov 13. PMID 41242336